CLINICAL TRIAL: NCT01657565
Title: Appendectomy in Children Performed by Residents in the Era of Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Nicolaj Markus Stilling, Doctor, Odense University Hospital
Other Study IDs: ED209; Appendectomy in children (Registry Identifier: NMS OUH)
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Intraabdominal Abscess; Wound Infection
Keywords: LOS; Ileus; Fever; reoperation
MeSH Terms: conditions — Wound Infection; Ileus; Fever

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- open appendectomy
- laparscopic appendectomy

SUMMARY:
Introduction: An increasing proportion of childhood appendicitis is treated with laparoscopic appendectomy (LA). The investigators wanted to elucidate the outcome of childhood appendicitis treated primarily by residents in a university hospital.

Material and methods: All children (age<16 years) treated surgically with appendectomy in our department between January 2006 and January 2011 were retrospectively identified. Readmission, reoperation or postoperative length of stay (LOS) exceeding five days were considered as non-satisfactory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age below 16 years. operated on suspicion of appendicitis

Exclusion Criteria:

* appendectomy for causes other than suspicion of appendicitis

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children 0-15 years of age having an appendectomy
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2006-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Surgical complications | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Stilling NM, Fristrup C, Gabers T, Qvist N, Rasmussen L. Acceptable outcome after laparoscopic appendectomy in children. Dan Med J. 2013 Jan;60(1):A4564. PMID 23340188